CLINICAL TRIAL: NCT04631523
Title: Investigation of the Relationship Between Internet Gaming Disorder and Reaction Time, Motor Dexterity, Neck Posture and Proprioception in Adolescents
Brief Title: Investigation of the Relationship Between Internet Gaming Disorder and Sensorimotor Functions in Adolescents
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aybike Senel, PT, MSc, Research Assistant, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 120
Record Dates: First submitted 2020-11-02; First posted 2020-11-17 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Internet Gaming Disorder
Keywords: internet gaming disorder; fine motor skills; adolescent; sensorimotor function
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IGD Group: The eligibility criteria were for IGD group as follows: being male in age between 10-18 years old; having accepted the research on a voluntary basis and signed the informed consent and being diagnosed with IGD according to DSM-5. Healthy adolescents in this study will be referred from a child and adolescent psychiatrist. All the following assessments will be applied this group for one time; Internet Addiction Scale, 9 Hole Peg Test, Ruler Drop Method, assessment of Forward Head Posture, evaluation of Joint Position Error of cervical region.
- Healthy Group: The eligibility criteria were for healthy group as follows: being male in age between 10-18 years old and having accepted the research on a voluntary basis and signed the informed consent. The adolescents with IGD in this study will be referred from a child and adolescent psychiatrist. All the following assessments will be applied this group for one time; Internet Addiction Scale, 9 Hole Peg Test, Ruler Drop Method, assessment of Forward Head Posture, evaluation of Joint Position Error of cervical region.

SUMMARY:
Using computer for long have been shown to cause vision problems, musculoskeletal pain particularly in neck, postural deviations, obesity and physical inactivity in several studies. The relation between obesity and physical activity, neck pain and postural deviations with altered sensorimotor function has been also shown with many studies. However, there were not enough study that assess sensorimotor congruence such as proprioception and reaction time in adolescents diagnosed with Internet Gaming Disorder (IGD). This study aimed to evaluate the proprioception and reaction time and investigate its relation with the relationship with neck pain, proprioception and reaction time in adolescents with IGD.

DETAILED DESCRIPTION:
The aim of this study is to evaluate reaction time, motor dexterity, cervical posture and proprioception and its relationship with Internet Gaming Disorder (IGD) in adolescents. It's anticipated that 60 adolescents aged between 10-18 years will be included to this study (30 healthy adolescent; 30 adolescent with IGD. After recording sociodemografic data of participants, age of starting to use the internet, the age of starting to play games on the internet, the time spent on the internet, the name and type of the game played will be questioned. The presence of musculoskeletal pain and its localization, if any, will be recorded. The severity of internet addiction will be assessed with Internet Addiction Scale, motor dexterity will be assessed with The 9 Hole Peg Test, reaction time of upper extremity will be assessed with Ruler Drop Method, the severity of forward head posture will be assessed with Cervical Range of Motion (CROM) device, and lastly, proprioception of cervical region will be assessed with Joint Position Error which will be evaluated CROM device. All parameters will be compared between healthy adolescents and adolescents with IGD.

ELIGIBILITY:
Inclusion Criteria:

For healthy group as follows:

* being male in age between 10-18 years old
* having accepted the research on a voluntary basis and signed the informed consent.

For the experimental group, being diagnosed with IGD according to DSM-5 is an additional criterion.

Exclusion Criteria:

* being diagnosed with psychotic, bipolar, or autism spectrum disorder
* the presence of mental retardation in the child or family that prevents answering the questions and following the instructions properly in clinical assessment
* Use of psychotropic drugs.

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will include 60 male adolescents diagnosed with Internet Gaming Disorder by the psychiatrist in Basaksehir Cam and Sakura City Hospital Child and Adolescent Psychiatry, Istanbul. The individuals who volunteers and meets the inclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Internet Addiction Scale | baseline
  It is a 20-itemed Likert type scale whose items are grading "Rarely", "Occasionally", "Often", "Most of the time" or "Always" with points of 1,2,3,4,5, respectively. The lowest score that can be obtained from the test is 20 and the highest score is 100. A score of 80 and above is an indicator of significant impairment in functionality and this group was defined as "internet addicted". Scores of "49 points and below" were defined as the "average internet user" who does not have any problems related to internet use in his life.

SECONDARY OUTCOMES:
9 Hole Peg Test | baseline
  The pegboard will be placed on table at midline of the body. The height of the table will be same at the participants' chest level. The participants will be asked to place the nine sticks into nine holes as quickly as possible and remove them immediately after finishing. The time will be begin on the first contact with the first stick and stopped last stick dropped.
Ruler Drop Method | baseline
  Ruler Drop Method will be used to assess reaction time. Participants will be made to sit with their dominant arm on table, elbow will be flexed at 90º and forearm will be mid-pronated. The ruler will be stabilized vertically by the examiner while the participants hold at the 5 cm with his/her web space (i.e. thumb and index finger). The participants will be asked to catch the ruler as fast as possible, after the ruler released from examiner's hand. The distance the ruler travelled from the starting point will be recorded as cm. This distance will be converted into time (sec) by using following formula "t =√(2d / g)".
Forward Head Posture | baseline
  The severity of forward heaad posture will assessed with CROM device according to CROM Procedure Manual. Participants will instructed to sit erect posture with spine away from the chair and feet flat on the floor. The horizontal bar with measured will be placed on the head, the vertical bar, whose lower end will be positioned over the spinal process of the 7th cervical vertebra (C7). After the resting point, where the vertical bar will be on, will be noted, the participants will be instructed to retract their heads as possible. The displacement in the sagittal plane will be recorded in cm.
Proprioception | baseline
  Joint position error (JPE) was measured to assess neck reposition sense of participants. For this test, the participants will be seated in chair with an erect posture, the examiner will stabilize the CROM device with the Velcro strap on participants head. They will be asked to focus a point on the wall as a feedback for neutral position. After the device will be calibrated to neutral position, the participants will perform an active left and right cervical rotation with eyes opened. This test will be repeated with eyes closed. The difference between reading values on the CROM device each side of rotation starting position and final position of the head (JPE) will be recorded as degree.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru KAYA MUTLU, PT, Assoc, Prof, Study Director — İstanbul University-Cerrahpaşa
Locations (1):
- İstanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)